CLINICAL TRIAL: NCT03348358
Title: How do Different Genres of Music Played During Labor Effect the Stress Level and the Obstetric and Perinatal Results?
Brief Title: Effect of Music on Stress and Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Yael Pasternak, Principal Investigator, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Music in delivery room
Record Dates: First submitted 2017-10-01; First posted 2017-11-20 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Stress; Delivery Problem for Fetus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Placebo Comparator): No music during labor
  Interventions: Behavioral: control
- Quiet music (Experimental): Women hearing quiet music during labor
  Interventions: Behavioral: quiet music
- Rhythmic music (Experimental): Women hearing rhythmic music during labor
  Interventions: Behavioral: Rhythmic music

INTERVENTIONS:
Behavioral: quiet music — playing quiet music during labor
  Arms: Quiet music
Behavioral: Rhythmic music — playing rhythmic music during labor
  Arms: Rhythmic music
Behavioral: control — No music during labor
  Arms: control

SUMMARY:
The purpose of this study is to randomize women to be exposed during labor to different genres of music and study the effect of each genre on the level of objective and subjective stress as manifested by salivary cortisol and personal stress questionnaires, respectively. Secondary outcomes to be examined are obstetric and perinatal outcomes

DETAILED DESCRIPTION:
For centuries, music has been known to have therapeutic effects on the body and the mind A large body of findings is related to the therapeutic potential of music in clinical settings, mainly among patients undergoing surgical and dental procedures, and also in other medical environments, such as intensive care, psychiatry, and geriatrics. Using music interventions in clinical settings was associated with reductions in negative effects in addition to objective stress and anxiety indices such as reduced heart rate, blood pressure, myocardial oxygen consumption, gastrointestinal function, anxiety, pain, and increased oxytocin levels.

One study found that women who listened to music before a cesarean section had a significant increase in positive emotions and a significant reduction in systolic blood pressure compared with a significant increase in diastolic blood pressure and respiratory rate in the control group. Li and Dong concluded in a different study, that preoperative music intervention can reduce anxiety and pain in women undergoing cesarean delivery.

Various studies examined the relation of music during labor to pain relief. One study found that the group of women going through music therapy had significantly lower pain, anxiety and a higher finger temperature during the latent phase of labor. One randomly assigned study found that women listened to soft music starting early in the active phase of labor had decreased sensation and distress of active labor pain. To date, no study examined the level of salivary cortisol while music is played at delivery room as an objective estimation of the stress level.

In addition to that, there is a lack of information regarding the effect of music during labor on the obstetric and perinatal outcomes.

Therefore, the purpose of this study is to randomize women to be exposed during labor to different genres of music and study the effect of each genre on the level of objective and subjective stress as manifested by salivary cortisol and personal stress questionnaire, respectively. Secondary outcomes to be examined are obstetric and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45
* single embryo
* term labor, >=37 weeks of gestation

Exclusion Criteria:

* multiple embryos
* Antepartum fetal death
* preterm delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Objective stress | An hour after administration to delivery room
  Stress as measured by saliva cortisol
Subjective stress | An hour after administration to delivery room
  Stress as measured by questionnaires

SECONDARY OUTCOMES:
Mode of delivery | through study completion, an average of 1 year
  Cesarean delivery/ vaginal delivery/ operative delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical center, Kfar Saba, Israel